CLINICAL TRIAL: NCT03250429
Title: Nasal and Peripheral Blood Biomarkers of CRS Patients Before and After Surgical Intervention
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Flight Attendant Medical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 17-1499
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Sinusitis, Chronic
MeSH Terms: conditions — Sinusitis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, urine, nasal lavage fluid, nasal epithelial lining fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRS subjects: CRS subjects who have sinus surgery
  Interventions: Procedure: Sinus surgery

INTERVENTIONS:
Procedure: Sinus surgery — Standard Clinical Sinus Surgery

SUMMARY:
To characterize inflammatory cells in the nose of patients with Chronic Rhinosinusitis (CRS) before and after sinus surgery.

DETAILED DESCRIPTION:
Rhinosinusitis (RS) is a heterogenous disease, with variable etiologies, manifestations, and progression. Generally, RS can be divided into acute, subacute, and chronic RS, depending on the symptoms and duration of the disease. Most commonly, acute RS is caused by a viral infection (viral RS), which starts in the nasal passages and progresses to inflammation of the sinuses. When this inflammation of the paranasal sinuses does not resolve and lasts for at least 12 weeks, the disorder is broadly defined as chronic RS (CRS), which is usually accompanied by bacterial infections. This inflammatory disease pathophysiology is further subdivided into CRS with (CRSwNP) and without (CRSsNP) nasal polyps. Recently, several studies aimed at phenotyping the diverse pathophysiology among patients suffering from CRS characterized subgroups based on the presence of inflammatory clusters. CRSsNP is marked by pro-inflammatory neutrophilic inflammation of the nasal mucosa and a nasal cytokine profile that is characterized by increased levels of TGFβ1 and IFNγ and low or undetectable levels of IL-5. In contrast, patients with CRSwNP demonstrate eosinophilic inflammation of the nasal mucosa, low levels of TGFβ1, but high levels of Th2/Th17-type cytokines such as IL-17 and IL-5, higher levels of eosinophil cationic protein (ECP) and mast cell tryptase, and lower levels of IL-10.

Currently biomarkers associated with physician diagnosed disease severity and patient-perceived quality of life impairments are lacking. Analysis of markers of inflammation in the nasal mucosa and peripheral blood leukocytes in combination with quality of life symptom scoring will enable us to identify biomarkers associated with CRS disease severity. This study will determine if biomarkers identified in the nasal mucosa and peripheral blood leukocytes correlate with physician diagnosed and patient-perceived disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed CRS with surgical requirement for treatment

Exclusion Criteria:

* Subjects with physician-diagnosed:
* cystic fibrosis,
* vasculitis,
* any type of nasal tumor
* receiving ongoing immunosuppressant therapy

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects who are patients at UNC Healthcare ENT clinics
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Inflammatory mediators in the nasal mucosa | Baseline (Pre-surgery), Post-surgery (approximately 12 weeks after surgery)
  Detection and analysis of inflammatory mediators previously characterized in CRS subgroups, including but not limited to Transforming growth factor beta 1 (TGFβ1), Interferon gamma (IFNγ), Interleukin 5 (IL-5), Interleukin 17 (IL-17), eosinophil cationic protein (ECP), mast cell tryptase, and Interleukin (IL-10) from the nasal mucosa.

SECONDARY OUTCOMES:
Change in Inflammatory mediators in the peripheral blood | Baseline (Pre-surgery), Post-surgery (approximately 12 weeks after surgery)
  Detection and analysis of inflammatory mediators previously characterized in CRS subgroups, including but not limited to TGFβ1, IFNγ, IL-5, IL-17, ECP, mast cell tryptase, and IL-10 from the peripheral blood.
Change in Rhinosinusitis Disability Index (RSDI) Scores | Baseline (Pre-surgery), Post-surgery (approximately 12 weeks after surgery)
  The RSDI is a disease-specific health-related quality of life instrument with 3 domains (physical, functional, and emotional impacts of rhinosinusitis) using a 5-point Likert scale ranging from 0 to 4 where 0 is "never" and 4 is "always a problem". Higher scores indicate more significant impact on quality of life.
Change in gene expression profile | Baseline (Pre-surgery), Post-surgery (approximately 12 weeks after surgery)
  Analyze cells for gene expression of inflammatory mediators including but not limited to TGFβ1, IFNγ, IL-5, IL-17, ECP, mast cell tryptase, and IL-10
Change in Nasal lavage fluid cell count | Baseline (Pre-surgery), Post-surgery (approximately 12 weeks after surgery)
  Count cell types present in nasal lavage fluid cells.

CONTACTS AND LOCATIONS:
Overall Officials: Ilona Jaspers, Ph.D., Principal Investigator — UNC SOM
Locations (1):
- Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No